CLINICAL TRIAL: NCT02975856
Title: Bioavailability of Table Red Wine and Young Port Red Wine Anthocyanins
Brief Title: Bioavailability of Red Wine Anthocyanins
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: REQUIMTE/LAQV, Departamento de Química e Bioquímica, FCUP (Unknown); Center for Health Technology and Services Research (Other); Vinoflavo (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: VINOFLAVO_02
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Anthocyanins; Bioavailability; Flavonoids; Port wine; Red wine

ARMS (2):
- Table Red Wine (Experimental): 250 ml Table Red Wine (12% ethanol)
  Interventions: Dietary Supplement: Table Red Wine
- Young Port Red Wine (Experimental): 150 ml Young Port Red Wine (20% ethanol)
  Interventions: Dietary Supplement: Young Port Red Wine

INTERVENTIONS:
Dietary Supplement: Table Red Wine
  Arms: Table Red Wine
Dietary Supplement: Young Port Red Wine
  Arms: Young Port Red Wine

SUMMARY:
The main aim of this study is to evaluate the bioavailability of table red wine and young Port red wine anthocyanins in healthy men.

DETAILED DESCRIPTION:
Anthocyanins (ANT) are water soluble pigments found in plants, flowers and fruits that are consumed as part of the human diet, many times in higher amounts than other flavonoid classes. Red wine is also an important source of anthocyanins, especially Mv3glc.

Several epidemiological studies have suggested that the consumption of anthocyanin-rich foods, including the moderate consumption of red wine, is positively associated with the prevention of cardiovascular heart disease.

It has become clear that the flavonoid bioactive forms in vivo are not necessarily those which occur in nature, but metabolites arising after absorption takes place.Therefore, studying the bioavailability of red wine ANT is very important to identify which metabolites (originated in vivo) can actually reach the target organs (and in which concentrations) and may be responsible for the postulated health benefits of red wine.

Intervention protocol:

Urine samples and peripheral venous blood (10 ml) will be collected from 10 h-fasting subjects. Afterwards, each volunteer will consume 250 ml of table red wine or 150 ml of young Port red wine and blood samples will be collected 15, 30, 60 and 120 min after wines ingestion. Another urine sample will be collected at 120 min.

Table red wine 12 % (250 ml) and young Port red wine 20 % (150 ml), two different food matrices rich in ANT, provided the same amount of ethanol (24 g of ethanol).

A thorough screening analysis for ANT will be performed in plasma and urine samples collected from the volunteers at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Age 18-65 years
* BMI < 25 kg/m2
* Willing and able to provide written consent

Exclusion Criteria:

* Subjects with current or previous CVD, diabetes or other severe chronic disease
* Subjects under prescription of any chronic medication
* Intake of red fruits or red wine in the last 24 h prior to the beginning of the intervention
* Subjects involved in any clinical or food study within the preceding month

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of anthocyanins and anthocyanins metabolites | At baseline and 15, 30, 60 and 120 minutes after wines consumption

SECONDARY OUTCOMES:
Urinary concentrations of anthocyanins and anthocyanins metabolites | At baseline and 120 minutes after wines consumption

CONTACTS AND LOCATIONS:
Overall Officials: Conceição Calhau, PhD, Principal Investigator — CINTESIS - Faculty of Medicine of University of Porto
Locations (1):
- CINTESIS - Faculty of Medicine of the University of Porto, Porto, Portugal